CLINICAL TRIAL: NCT02397967
Title: Neuropsychological Characterisation of Cognitive Deficits Involved in Reading Disability in Children With NF1
Brief Title: Reading Disability in Children With NF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 08 113 01
Record Dates: First submitted 2015-03-13; First posted 2015-03-25 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Neurofibromatosis Type 1
Keywords: NF1; children; reading disabilities
MeSH Terms: conditions — Neurofibromatosis 1; Dyslexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Children NF1 (Experimental): Children diagnosed with NF1 according the NIH criteria Neuropsychological assessments
  Interventions: Other: Neuropsychological assessments
- Control group (Placebo Comparator): Control group children without NF1 with the same reading level Neuropsychological assessments
  Interventions: Other: Neuropsychological assessments

INTERVENTIONS:
Other: Neuropsychological assessments — Neuropsychological assessments:
  Intelligence Quotient (WISC-IV)
  Reading tests (reading accuracy, reading speed, reading comprehension and strategy):
  Alouette test, Lobrot test, Odedys test. Visio-spatial skill (JLO, Thurston, Corsi tests) Attention (CPT 2, CBCL) Receptive oral language (EVIP)

SUMMARY:
A national, multicenter, randomized, transverse clinical trial, estimating the existence of phonological deficits in children with NF1 children compared with control children without NF1 with the same reading level.

DETAILED DESCRIPTION:
To determine the phonological and visio -spatial performances at the NF1 children.

ELIGIBILITY:
Inclusion Criteria:

* Age included between 8 and 12 years
* Child presenting a type 1 neurofibromatosis according to 2 criteria in the following criteria list :

  * At least 6 café au lait spots
  * 2 or more neurofibromas or 1 plexiform neurofibroma
  * axillary or inguinal freckling
  * 1 optic nerf glioma
  * 2 or more Lisch nodules
  * 1 osseous lesion as sphenoid dysplasia or thinning of the long bone cortex with or without pseudoarthrosis
  * 1 A first degree relative (parent, sibling, or offspring) with NF1 by the above criteria
* Membership in a national insurance
* Consent of the child and the parents

Exclusion Criteria:

* Mental retardation (QI T < 70)
* Treated or untreated epilepsy
* Visual deficit (visual Acuteness < 4/10
* Presence of a symptomatic optic glioma
* Presence of a brain tumor.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2009-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Phonological deficits evaluated by the metaphonological capabilities including a subtraction test and phonemic Acronym test and memory capacity with phonological phonological memory test. | 24 hours
  Evaluate whether there is a specificity of phonological deficits in children with NF1 compared with a population of children with the same age and same reading level, taking into account the intellectual level.

SECONDARY OUTCOMES:
Visual-perceptual performance established from three tests: Test of Identical Forms (Thurstone), Judgment Test of orientation Lines (Benton) and global and partial deferral Tasks (S Valdois). | 24 hours
  Studying the correlations between phonological deficits and visio-spatial and literacy skills.

CONTACTS AND LOCATIONS:
Overall Officials: Yves CHAIX, Professor, Principal Investigator
Locations (6):
- France (6):
  - Hopital femme-mére-enfant, Hospices civils de lyon, Lyon
  - Hôpital Gui de Chauliac, Montpellier
  - CHU Hôtel-Dieu, Clinic of Dermatology, Nantes
  - AP-HP Hopital Armand Trousseau, Paris
  - Hôpital des Enfants, Toulouse
  - Hopital Gatien de Clocheville, Tours

REFERENCES:
- [Derived] Biotteau M, Tournay E, Baudou E, Destarac S, Iannuzzi S, Faure-Marie N, Castelnau P, Schweitzer E, Rodriguez D, Kemlin I, Dorison N, Rivier F, Carneiro M, Preclaire E, Barbarot S, Lauwers-Cances V, Chaix Y. Reading Comprehension Impairment in Children With Neurofibromatosis Type 1 (NF1): The Need of Multimodal Assessment of Attention. J Child Neurol. 2021 Jul;36(8):625-634. doi: 10.1177/0883073820981270. Epub 2021 Jan 28. PMID 33507832